CLINICAL TRIAL: NCT05008185
Title: Regenerative Peripheral Nerve Interfaces to Treat Painful Digit and Hand Neuromas After Amputation: A Prospective Observational Trial"
Brief Title: Regenerative Peripheral Nerve Interfaces to Treat Painful Digit and Hand Neuromas After Amputation
Status: Recruiting | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00049513
Record Dates: First submitted 2021-07-28; First posted 2021-08-17 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Neuroma
Keywords: Neuroma; Neuroma Pain; Finger Amputation; Hand Amputation
MeSH Terms: conditions — Neuroma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regenerative Peripheral Nerve Interface: symptomatic neuroma is excised, and the end of the peripheral nerve is implanted into a small denervated free muscle graft harvested from the patient
  Interventions: Procedure: Regenerative Peripheral Nerve Interface (RPNI) surgery
- Traction Neurectomy: simple excision and traction neurectomy
  Interventions: Procedure: Traction Neurectomy

INTERVENTIONS:
Procedure: Regenerative Peripheral Nerve Interface (RPNI) surgery — Surgeons will perform neuroma resection and RPNI creation using a free muscle graft from the brachioradialis muscle harvested through a small separate incision
  Groups: Regenerative Peripheral Nerve Interface
Procedure: Traction Neurectomy — Surgeons will perform neuroma resection and traction neurectomy,
  Groups: Traction Neurectomy

SUMMARY:
This study is being done to demonstrate the effectiveness of Regenerative Peripheral Nerve Interfaces (RPNI) surgery in treating symptomatic neuromas of the hand and digits following amputation compared to standard of care using a Prospective, Observational Trial

DETAILED DESCRIPTION:
This will be a prospective observational study that seeks to provide a comprehensive assessment of the outcomes after RPNI surgery compared to standard of care by utilizing multiple established and validated patient-reported outcomes measures, carefully tracking pre- and post-operative pain regimens, and performing functional and physiologic tests.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* History of unilateral digit, multiple digit, or partial hand amputation
* Discrete neuroma pain on clinical exam
* Following standard of care (SOC), confirmation through a local block and/or ultrasound imaging will be performed if indicated
* Must be seen by a hand therapist for at least 6-week trial of desensitization therapy

Exclusion Criteria:

* Patients with previous surgical treatment for symptomatic neuromas of the digits or hand
* Patients with other major injuries more proximal in the ipsilateral extremity that cause chronic pain or functional loss
* women pregnant at time of enrollment
* prisoners
* adults who are unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with a history of digit, multi-digit or partial hand amputation. Patients must have discrete neuroma pain on clinical exam.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System - Pain Interference (PROMIS-PI) | Assessing change from Baseline to 1 week, 1 month, 3 months and 6 months
  PROMIS Pain Interference (PROMIS-PI) scale measures the extent to which pain hinders an individual's engagement with physical, mental, cognitive, emotional, recreational, and social activities over the past 7 days answering each questions with a response of not at all, a little bit, somewhat, quite a bit, and very much with not at all being the best and very much the worst.
Short-form McGill Pain Questionnaire (SF-MPQ-2) | Assessing change from Baseline to 1 week, 1 month, 3 months and 6 months
  theShort-form McGill Pain Questionnaire (SF-MPQ-2) measures 24 different qualities of pain and related symptoms using the intensity of pain and related symptoms felt during the past week on 0 to 10 scale, with 0 being no pain and 10 being the worst pain .
PROMIS Global Health (GH) v1.2 | Assessing change from Baseline to 1 week, 1 month, 3 months and 6 months
  The Global Health Questionnaire contains 10 questions (7 general and 3 about the last 7 days). First 7 questions use a scale of excellent, very good, good, fair, and poor, poor being the worst with excellent being the best. The other three questions use different scales such as; never rarely, sometimes, often or always with never being the best and always being the worst; as well as none, mild, moderate, severe, very severe with none being the best and very severe being the worst; finally pain rating numbered 0-10 with 0 being no pain and 10 being the worst pain imaginable.
Patient Health Questionnaire (PHQ-9), | Assessing change from Baseline to 1 week, 1 month, 3 months and 6 months
  The PHQ-9 form is a brief, self-administered questionnaire that assesses depression symptoms over the last 2 weeks consisting of 10 questions. 9 will be answered on a scale of 0-3 with 0 being the best and 3 bing the worst. The last question will use a response of not difficult at all, somewhat difficult, very difficult, and extremely difficult with not difficult at all being the best and extremely difficult being the worst.
Generalized Anxiety Disorder measure (GAD-7), | Assessing change from Baseline to 1 week, 1 month, 3 months and 6 months
  Generalized Anxiety Disorder measure (GAD-7) is a screening tool and severity measure for generalised anxiety disorder (GAD) over the past 2 weeks consisting of 7 questions answered on a scale of 0-3 with 0 being the best and 3 being the worst.
PC-PTSD-5 | Assessing change from Baseline to 1 week, 1 month, 3 months and 6 months
  The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) is a 5-item screening tool with 'Yes/No" answers designed to identify individuals with probable PTSD. Yes" answers represent the worst and "no" represents the best.

SECONDARY OUTCOMES:
PROMIS UpperExtremity (UE) | Assessing change from Baseline to 1 week, 1 month, 3 months and 6 months
  PROMIS UpperExtremity (UE) is designed to evaluate upper extremity function using a scale of 1-5 with 5 being the best possible answer and 1 being the worst.
Brief Michigan Hand Outcomes Questionnaire (bMHQ) | Assessing change from Baseline to 1 week, 1 month, 3 months and 6 months
  The Brief Michigan Hand Outcomes Questionnaire (bMHQ) evaluates six upper extremity domains of function, activities of daily living(ADLs), aesthetics, performance,pain,and satisfaction using a scale of 1-5 with 5 being the best possible answer and 1 being the worst.
Grip Strength | Assessing change from Baseline to 1 month, 3 months and 6 months
  A standard dynamometer will be used to evaluate grip strength
Pinch Strength -Key and Three-point | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate key pinch (thumb to radial border of index) and three-point pinch (index, middle, and thumb tips) strength.
Range of Motion | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate active and passive range of motion of all joints in the affected extremity proximal to the amputation stump, total active and passive range of motion of all unaffected digits on the ipsilateral hand, and total active motion of fall digits and wrist on the contralateral hand as an internal control
Fine Motor Function - 9-Hole Peg Test (9HPT) | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate timed exercise during which nine relatively small pegs are picked up, one at a time, and put into nine corresponding holes. The pegs are then removed from the holes (one at a time) and placed back in the starting bin.
FunctionalTask Testing - Lifting boxes | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate whether the participant is able to perform the task, grip that was used, maximum weight used, and any compensatory findings. Subjects will be asked their pain level during each lift using a 10-point numerical scale
Functional Task Testing - Carrying Boxes | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate whether the participant is able to perform the task, grip that was used, maximum weight used, and any compensatory findings. Subjects will be asked their pain level during each lift using a 10-point numerical scale
Functional Task Testing - Push/Pull sled | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate whether the participant is able to perform the task, grip that was used, maximum weight used, and any compensatory findings. Subjects will be asked their pain level during each lift using a 10-point numerical scale
Functional Task Testing - Hammer | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate tolerance for vibration and grip to perform a hammer task using
Functional Task Testing - Vice Grip | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate vice grip Strength with all available digits using the Baltimore Therapeutic Equipment (BTE) PrimusRS work simulator.
Functional Task Testing - Gear Shifting | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate ability to grip, push and pull gear shift with all available digits using the Baltimore Therapeutic Equipment (BTE) PrimusRS work simulator
Functional Task Testing - Weapon Recoil | Assessing change from Baseline to 1 month, 3 months and 6 months
  Evaluate the ability to preform this simulated task using the Baltimore Therapeutic Equipment (BTE) PrimusRS work simulator

CONTACTS AND LOCATIONS:
Overall Officials: Aviram M Giladi, MS, MD, Principal Investigator — Medstar Union Memorial Hospital
Locations (2):
- United States (2):
  - The Curtis National Hand Center at Medstar Union Memorial Hospital, Baltimore, Maryland
  - University of Michigan Plastic Surgery, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woo SL, Kung TA, Brown DL, Leonard JA, Kelly BM, Cederna PS. Regenerative Peripheral Nerve Interfaces for the Treatment of Postamputation Neuroma Pain: A Pilot Study. Plast Reconstr Surg Glob Open. 2016 Dec 27;4(12):e1038. doi: 10.1097/GOX.0000000000001038. eCollection 2016 Dec. PMID 28293490
- [Background] Urbanchek MG, Kung TA, Frost CM, Martin DC, Larkin LM, Wollstein A, Cederna PS. Development of a Regenerative Peripheral Nerve Interface for Control of a Neuroprosthetic Limb. Biomed Res Int. 2016;2016:5726730. doi: 10.1155/2016/5726730. Epub 2016 May 17. PMID 27294122
- [Background] Santosa KB, Oliver JD, Cederna PS, Kung TA. Regenerative Peripheral Nerve Interfaces for Prevention and Management of Neuromas. Clin Plast Surg. 2020 Apr;47(2):311-321. doi: 10.1016/j.cps.2020.01.004. Epub 2020 Feb 1. PMID 32115057
- [Background] Kemp SW, Cederna PS, Midha R. Comparative outcome measures in peripheral regeneration studies. Exp Neurol. 2017 Jan;287(Pt 3):348-357. doi: 10.1016/j.expneurol.2016.04.011. Epub 2016 Apr 17. PMID 27094121
- [Background] Ursu DC, Urbanchek MG, Nedic A, Cederna PS, Gillespie RB. In vivo characterization of regenerative peripheral nerve interface function. J Neural Eng. 2016 Apr;13(2):026012. doi: 10.1088/1741-2560/13/2/026012. Epub 2016 Feb 9. PMID 26859115
- [Background] Giladi AM, McGlinn EP, Shauver MJ, Voice TP, Chung KC. Measuring outcomes and determining long-term disability after revision amputation for treatment of traumatic finger and thumb amputation injuries. Plast Reconstr Surg. 2014 Nov;134(5):746e-755e. doi: 10.1097/PRS.0000000000000591. PMID 25347649
- [Background] Langhals NB, Woo SL, Moon JD, Larson JV, Leach MK, Cederna PS, Urbanchek MG. Electrically stimulated signals from a long-term Regenerative Peripheral Nerve Interface. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1989-92. doi: 10.1109/EMBC.2014.6944004. PMID 25570372
- [Background] Frost CM, Cederna PS, Martin DC, Shim BS, Urbanchek MG. Decellular biological scaffold polymerized with PEDOT for improving peripheral nerve interface charge transfer. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:422-5. doi: 10.1109/EMBC.2014.6943618. PMID 25569986
- [Background] Woo SL, Urbanchek MG, Cederna PS, Langhals NB. Revisiting nonvascularized partial muscle grafts: a novel use for prosthetic control. Plast Reconstr Surg. 2014 Aug;134(2):344e-346e. doi: 10.1097/PRS.0000000000000317. No abstract available. PMID 25068369
- [Background] Kung TA, Langhals NB, Martin DC, Johnson PJ, Cederna PS, Urbanchek MG. Regenerative peripheral nerve interface viability and signal transduction with an implanted electrode. Plast Reconstr Surg. 2014 Jun;133(6):1380-1394. doi: 10.1097/PRS.0000000000000168. PMID 24867721
- [Background] Kung TA, Bueno RA, Alkhalefah GK, Langhals NB, Urbanchek MG, Cederna PS. Innovations in prosthetic interfaces for the upper extremity. Plast Reconstr Surg. 2013 Dec;132(6):1515-1523. doi: 10.1097/PRS.0b013e3182a97e5f. PMID 24281580
- [Background] Hooper RC, Cederna PS, Brown DL, Haase SC, Waljee JF, Egeland BM, Kelley BP, Kung TA. Regenerative Peripheral Nerve Interfaces for the Management of Symptomatic Hand and Digital Neuromas. Plast Reconstr Surg Glob Open. 2020 Jun 4;8(6):e2792. doi: 10.1097/GOX.0000000000002792. eCollection 2020 Jun. PMID 32766027
- [Background] Svientek SR, Ursu DC, Cederna PS, Kemp SWP. Fabrication of the Composite Regenerative Peripheral Nerve Interface (C-RPNI) in the Adult Rat. J Vis Exp. 2020 Feb 25;(156):10.3791/60841. doi: 10.3791/60841. PMID 32176203
- [Background] Vu PP, Vaskov AK, Irwin ZT, Henning PT, Lueders DR, Laidlaw AT, Davis AJ, Nu CS, Gates DH, Gillespie RB, Kemp SWP, Kung TA, Chestek CA, Cederna PS. A regenerative peripheral nerve interface allows real-time control of an artificial hand in upper limb amputees. Sci Transl Med. 2020 Mar 4;12(533):eaay2857. doi: 10.1126/scitranslmed.aay2857. PMID 32132217
- [Background] Frost CM, Ursu DC, Flattery SM, Nedic A, Hassett CA, Moon JD, Buchanan PJ, Brent Gillespie R, Kung TA, Kemp SWP, Cederna PS, Urbanchek MG. Regenerative peripheral nerve interfaces for real-time, proportional control of a Neuroprosthetic hand. J Neuroeng Rehabil. 2018 Nov 20;15(1):108. doi: 10.1186/s12984-018-0452-1. PMID 30458876
- [Background] Vu PP, Irwin ZT, Bullard AJ, Ambani SW, Sando IC, Urbanchek MG, Cederna PS, Chestek CA. Closed-Loop Continuous Hand Control via Chronic Recording of Regenerative Peripheral Nerve Interfaces. IEEE Trans Neural Syst Rehabil Eng. 2018 Feb;26(2):515-526. doi: 10.1109/TNSRE.2017.2772961. PMID 29432117
- [Background] Ursu D, Nedic A, Urbanchek M, Cederna P, Gillespie RB. Adjacent regenerative peripheral nerve interfaces produce phase-antagonist signals during voluntary walking in rats. J Neuroeng Rehabil. 2017 Apr 24;14(1):33. doi: 10.1186/s12984-017-0243-0. PMID 28438166
- [Background] Hart SE, Kung TA. Novel Approaches to Reduce Symptomatic Neuroma Pain After Limb Amputation. Curr Phys Med Rehabil Rep. 2020 Jun 16;(8):83-91.